CLINICAL TRIAL: NCT03505970
Title: Blood and Muscle Responses to Sodium Bicarbonate Supplementation and Subsequent Exercise Performance
Brief Title: Blood, Muscle and Exercise Responses to Sodium Bicarbonate Supplementation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: SB_BloodMuscle
Record Dates: First submitted 2018-03-31; First posted 2018-04-23 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Sports Nutritional Physiological Phenomena
Keywords: Physiological Phenomena
MeSH Terms: interventions — Sodium Bicarbonate; maltodextrin

STUDY DESIGN:
Intervention Model Description: Double-blind crossover
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium bicarbonate (Experimental): 0.3 g∙kg-1body mass of sodium bicarbonate
  Interventions: Dietary Supplement: Sodium bicarbonate
- Placebo (Placebo Comparator): Individuals will ingest 0.3 g/kg maltodextrin before undergoing exercise
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Sodium bicarbonate — Sodium bicarbonate in powder form ingested in gelatine capsules. This leads to an increase bicarbonate concentration in blood, increasing buffering capacity which may lead to improvements in exercise
  Arms: Sodium bicarbonate
Dietary Supplement: Maltodextrin — Maltodextrin will be used as a placebo as it will not lead to any increases in circulating bicarbonate and, at this dose, will not likely have any physiological effect.
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the changes in activity of transporters of H+ (monocarboxylate transporters; MCT1, MCT4, NHE) following sodium bicarbonate supplementation and subsequent exercise performance. Fifteen healthy men (age 18-35 years) will be invited to attend the laboratory on five separate visits to a randomized, double-blind, placebo-controlled study. Participants will be supplemented with a 0.3 g/kg dose of sodium bicarbonate or placebo (Analytical Pharmacy, Brazil) in opaque gelatin capsules. One hour after supplementation they will perform a 1-km time trial and every 10 minutes a blood sample will be collected. A muscle biopsy will be taken prior to supplementation, immediately prior to exercise, and immediately post-exercise. A questionnaire will be also used to evaluate the side-effects associated with sodium bicarbonate supplementation. Muscle and blood samples will be analysed for acidity and H+ and muscle samples will be analysed for H+ transporters (MCT1, MCT4, NHE).

ELIGIBILITY:
Inclusion Criteria:

* Healthy males

Exclusion Criteria:

* Smokers
* Chronic disease
* Prior or current use of steroids
* Use of creatine in the last 6 months
* Use of beta-alanine in the last 6 months

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
H+ transporter activity | 5 minutes Post-exercise
  Change in activity of transporters related to H+

SECONDARY OUTCOMES:
Exercise performance | 1 hour Post-supplementation
  Change in 1 km cycling time-trial performance